CLINICAL TRIAL: NCT06351098
Title: Longitudinal Investigation of Sleep, Memory, and Brain Development Across the Nap Transition
Acronym: HSR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Tracy Riggins, Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024579
Record Dates: First submitted 2024-03-15; First posted 2024-04-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Memory
Keywords: Sleep; Brain development

STUDY DESIGN:
Intervention Model Description: Memory will be assessed using the Mnemonic Similarity Task (MST), before and after nap/wake and overnight sleep. The specific variable of interest is the lure discrimination index, which refers to the probability of "Similar" responses to lure items minus the probability of "Similar" responses given to foils.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nap (Experimental): Children are nap promoted
  Interventions: Behavioral: nap

INTERVENTIONS:
Behavioral: nap — Children are nap promoted

SUMMARY:
To examine the relations between sleep (nap transitions, sleep physiology), memory, and brain development longitudinally, the researchers will assess n=180 children (in order to acquire n=152 usable data sets) who are 36-54 months of age and habitual nappers at enrollment. In each wave, the researchers will assess memory, memory change over a nap and equivalent waking interval, sleep physiology of the nap, and brain structure and function (using Magnetic Resonance Imagining or MRI). Additionally, overnight sleep physiology will be assessed in all participants. Waves will take place approximately every 6 months. For all children, three waves will be collected. With these data, the researchers will address the following aims:

* Examine neural markers that predict the sleep transition (Aim 1);
* Examine changes in sleep-dependent memory processing (mnemonic discrimination) over both nap and overnight sleep intervals, across the sleep transition (Aim 2);
* Examine changes in sleep microstructure in both nap and overnight sleep across the sleep transition (Aim 3)
* Examine interrelations among brain, memory and sleep microstructure across the sleep transition (Aim 4)

DETAILED DESCRIPTION:
Child participants will be recruited from databases maintained at each university (see Human Subjects). Initially, parent-report will determine whether the child qualifies as a habitual napper, which will later be confirmed by actigraphy. In each wave, participants will then complete 3 sessions, 3-7 days apart. The first two sessions will consist of nap or wake promotion (counter-balanced, separated by one week) and memory assessments. The third session will consist of a visit to the university for the MRI scan. All of the participants will also have overnight sleep and overnight sleep-dependent memory consolidation assessed on the evenings following the nap/wake sessions. An Actiwatch watch will be given to the participant at the beginning of the first wave. Instructions will be included describing how to put the watch on the child and that the watch should be worn as often as possible. Nap and wake sessions will begin 30 mins prior to the child's typical nap time (if habitual nappers) or approximately 12:30 pm (non-habitual nappers). First, children will complete the encoding and immediate retrieval phases of the mnemonic similarity task. Subsequently, children will either be nap- or wake-promoted. Polysomnography (PSG) will be applied in the nap condition, but timing will be equated in the wake condition. Thirty-minutes following wake (or approximately 3:30 pm for those in the wake group), children will complete the delayed retrieval phase of the mnemonic similarity task.

Participants at both testing sites will also have overnight sleep and memory assessed after the nap and wake sessions. Experimenters will arrive at the participant's house about 30 mins prior the child's typical bedtime. The child will encode a new set of stimuli and complete the immediate retrieval phase of the mnemonic discrimination task. Subsequently, the child will be fitted with PSG. Parents are given instructions on placement of the PSG amplifier during the night and how to remove in the electrodes in the morning. Experimenters will return in the morning to retrieve the equipment and obtain the delayed retrieval phase of the mnemonic similarity task. Approximately 3-7 days after the second visit, children will complete the MRI session. The researchers will attempt to obtain MRI scans in the morning to avoid confounds with nap status. The Actiwatch will also be collected in this session. Children will then be fitted with the Fitbit to wear as often as possible between testing waves. These procedures will be repeated every 6 months for 2-3 waves.

ELIGIBILITY:
Inclusion Criteria:

1. 36-60 months at the time of enrollment
2. must be a habitual napper (defined as napping 5 or more days/week on average for the past month)
3. must sleep independently (not bedsharing; in order to maintain consistent sleep not interrupted by others)

Exclusion Criteria:

1. diagnosis of any sleep disorder (other than mild parasomnia which is routine at this age) past or present (Child's Sleep Habit Questionnaire)
2. current use of psychotropic or sleep-altering medications (Developmental, Health, and Environment Questionnaire)
3. traveling beyond 1 time zone within 1 month prior to testing (phone screening)
4. fever or symptoms of respiratory illness at the time of testing (phone screening)
5. physical handicap which interferes with assessments (vision, hearing impairment; phone screening)
6. diagnosed developmental disability (Developmental, Health, and Environment Questionnaire)
7. history of neurological injury such as history of seizures, brain tumor, or stroke (phone screening)
8. presence of metal in the body (e.g., implant of any form) or other contraindication for MRI (e.g., claustrophobia, which is rare at this age).
9. external influences on nap habits (e.g., inability to nap due to school or caregiver schedule or interfering activities during a typical naptime) including if the child will enroll in full-day kindergarten by the end of the study. Caregivers will also be queried for the presence of interfering activities throughout enrollment (e.g., ecological momentary assessment (or EMA), sleep diaries at each wave).

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Memory | across the nap period, approximately 2.5 hours
  Memory will be assessed using the Mnemonic Similarity Task (MST), before and after nap/wake and overnight sleep. The specific variable of interest is the lure discrimination index, which refers to the probability of "Similar" responses to lure items minus the probability of "Similar" responses given to foils.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, College Park, Maryland
  - University of Massachusetts, Amherst, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected through the proposed work will be made available to researchers pursuant to the Policies of NIH and the University of Maryland. Access to data will be granted upon request to qualified academic investigators for non-commercial research. Research resources generated with funds from this grant will be freely distributed, as available, to qualified academic investigators for noncommercial research upon request. Finally, following publication, raw MRI and PSG data will also be made available on the National Sleep Research Resource (NSRR), which is supported by the National Heart, Lung, and Blood Institute. The NSRR offers access free-of-charge to collections of de-identified physiological signals and clinical data elements from well-characterized research cohorts and clinical trials. If MRI data prove difficult to upload to NSRR, we will work with NHLBI Program to identify a supplemental or additional repository for the MRI data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available following publication.
Access Criteria: Data will be made available to researchers pursuant to the Policies of NIH and the University of Maryland.